CLINICAL TRIAL: NCT01527526
Title: Prospective Study for Evaluation of the Insulin Resistance, Lipid Metabolism and Sub Clinical Cardiovascular Disease in Women Who Initiate the Depot-medroxyprogesterone Acetate (DMPA) Contraceptive Method With in Follow-up for Two Years
Brief Title: Depot-medroxyprogesterone Acetate (DMPA) Contraceptive Method and Metabolism
Acronym: DMPA
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luis Bahamondes, MD Medical Doctor, University of Campinas, Brazil
Other Study IDs: 09/2011/PC
Record Dates: First submitted 2011-11-16; First posted 2012-02-07 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Insulin Resistance; Cardiovascular Disease; Bone Loss; Eating Disorders; Thrombosis
Keywords: DMPA; insulin resistance; cardiovascular disease; BMI; weight gain; thrombosis
MeSH Terms: conditions — Insulin Resistance; Cardiovascular Diseases; Bone Diseases, Metabolic; Feeding and Eating Disorders; Thrombosis; Weight Gain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for determination of lipid profile, insulin, glucose, coagulation factors, neuropeptide Y and factors related to bone mineral density.
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective:

The purpose of this study is to determine the etiology of the weight increase in Depot-medroxyprogesterone Acetate (DMPA) users.

Method:

Prospective study with 100 women, aged 18-40 years old and BMI < 30kg/m², paired with users of a non hormonal method follow for two years. Will be included only women who never used DMPA. There will be evaluated habit, blood pressure, anthropometric measure, distribution of corporal fat, lipids profile and glycemia parameters every six months. Thirty women and their control group will performed a euglycemic-hyperinsulinemic clamp to evaluate the resistance of insulin, adiponectin,neuropeptide Y, apolipoprotein A/B and arterial evaluation with ultrasound, intimal and media measure. Anova analysis for repeated samples. The metabolic alterations should elucidate the etiology, and the beginning of the sub clinical cardiovascular disease should be shown/discarded with the arterial evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* new users of DMPA
* BMI<30kg/m²

Exclusion Criteria:

* diabetes mellitus and 2 present or fasting glucose> 100mg/dl and / or blood glucose> 140mg/dl after ingestion of 75mg of oral glucose
* first-degree relatives with diabetes mellitus
* period of lactation
* hypertension, with or without treatment
* hyper and hypothyroidism
* chronic renal failure
* transplant of any organ
* women using drugs that may be related to weight gain and / or development of insulin resistance and chronic use of corticosteroids, antipsychotics, statins, and thiazide,
* hirsutism and/or hyperandrogenism
* polycystic Ovary Syndrome (PCOS)
* women with acanthosis nigricans
* women who have used depoprovera at some point in their reproductive lives,
* women who have performed bariatric surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Will be included women new-users DMPA, looking for the clinic's family planning FCM-UNICAMP, from primary care centers in Campinas, São Paulo, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 12 months
  insulin resistance diagnosed by hyperinsulinemic-euglycemic clamp at 0 and 12 months

SECONDARY OUTCOMES:
weight gain | 12 months
  other arm of the study
eating disorder | 12 months
  other arm of the study
loss of bone mass | 12 months
  other arm of the study
changes in clotting factors | 12 months
  other arm of the study

CONTACTS AND LOCATIONS:
Overall Officials: Luis Bahamondes, M.D., Principal Investigator — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Modesto W, Bahamondes MV, Silva dos Santos P, Fernandes A, Dal'Ava N, Bahamondes L. Exploratory study of the effect of lifestyle counselling on bone mineral density and body composition in users of the contraceptive depot-medroxyprogesterone acetate. Eur J Contracept Reprod Health Care. 2014 Aug;19(4):244-9. doi: 10.3109/13625187.2014.924098. Epub 2014 Jun 13. PMID 24923792